CLINICAL TRIAL: NCT06600516
Title: Minimal Intervention Necessary for Change: a Pilot Randomized Clinical Trial Modifying Cognitive Behavioral Therapy for Insomnia to Improve Sleep and Cognitive Function
Brief Title: Assessing Modified CBTi in Adults with Insomnia Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2024-124
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insomnia Disorder; Cognitive Functioning
Keywords: Modified CBTi; Adults; Insomnia Disorder; Cognitive Functioning
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Pilot randomized clinical trial with 4 treatment groups: stimulus control, sleep restriction, sleep compression, waitlist control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stimulus Control (Active Comparator): Stimulus control.45 People with insomnia may fail to associate the bedroom with sleep, and instead may associate it with worrying, planning, or recreation. Stimulus control includes the following instructions: (1) go to bed only when sleepy; (2) only use your bed or bedroom for sleep (or sex); (3) if you do not fall asleep quickly (i.e., 15 minutes), leave the bed, do something in another room, and return to bed only when you feel a strong sleep urge; (4) if you do not fall asleep quickly upon returning to bed, repeat instruction 3; (5) use your alarm to awaken at the same time every morning regardless of duration of sleep obtained; and (6) do not take long naps.
  Interventions: Behavioral: CBTi: Stimulus Control Core
- Sleep Restriction (Active Comparator): Sleep restriction.46 People with insomnia often spend too much time awake in bed. Sleep restriction modifies the participant's sleep window so total time in bed is no more than 30 minutes beyond their average total sleep time to consolidate sleep, thus improving depth, continuity, and consistency. As the participant's sleep efficiency improves with treatment (i.e., the percentage of total time spent asleep within the sleep window), their sleep window is also increased. However, the shortened sleep window often causes increased anxiety.
  Interventions: Behavioral: CBTi: Sleep Restriction Core
- Sleep Compression (Active Comparator): Sleep compression.47,48 Sleep compression encourages time-in-bed restrictions. Unlike sleep restriction, sleep compression allows a gradual reduction in time-in-bed over the course of multiple weeks. Typically, average total sleep time and total time in bed values are calculated from one or more weeks of daily sleep diaries. The difference between these two values is then divided by the number of weeks remaining and the allotted time in bed duration is compressed by this calculated value weekly, by delaying bedtime or advancing wake time.
  Interventions: Behavioral: CBTi: Sleep Compression Core
- Waitlist Control (No Intervention): Waitlist Control. Those randomly assigned to the WLC group will be told that they must wait 4 weeks for treatment, which is a fraction of the typical wait period in routine clinical care. During this time the participants are asked to maintain their regular schedule. At the end of 4 weeks, they will complete the baseline assessments again, which will serve as the post-waitlist assessment and then scheduled with a clinician to receive CBTi.

INTERVENTIONS:
Behavioral: CBTi: Stimulus Control Core — Stimulus control.45 People with insomnia may fail to associate the bedroom with sleep, and instead may associate it with worrying, planning, or recreation. Stimulus control includes the following instructions: (1) go to bed only when sleepy; (2) only use your bed or bedroom for sleep (or sex); (3) if you do not fall asleep quickly (i.e., 15 minutes), leave the bed, do something in another room, and return to bed only when you feel a strong sleep urge; (4) if you do not fall asleep quickly upon returning to bed, repeat instruction 3; (5) use your alarm to awaken at the same time every morning regardless of duration of sleep obtained; and (6) do not take long naps.
  Arms: Stimulus Control
Behavioral: CBTi: Sleep Restriction Core — Sleep restriction.46 People with insomnia often spend too much time awake in bed. Sleep restriction modifies the participant's sleep window so total time in bed is no more than 30 minutes beyond their average total sleep time to consolidate sleep, thus improving depth, continuity, and consistency. As the participant's sleep efficiency improves with treatment (i.e., the percentage of total time spent asleep within the sleep window), their sleep window is also increased. However, the shortened sleep window often causes increased anxiety.
  Arms: Sleep Restriction
Behavioral: CBTi: Sleep Compression Core — Sleep compression.47,48 Sleep compression encourages time-in-bed restrictions. Unlike sleep restriction, sleep compression allows a gradual reduction in time-in-bed over the course of multiple weeks. Typically, average total sleep time and total time in bed values are calculated from one or more weeks of daily sleep diaries. The difference between these two values is then divided by the number of weeks remaining and the allotted time in bed duration is compressed by this calculated value weekly, by delaying bedtime or advancing wake time.
  Arms: Sleep Compression

SUMMARY:
Sleep is a biological need, crucial for maintaining overall health and resiliency. Sleep disorders disrupt this normal functioning. Insomnia disorder is the most prevalent sleep disorder and yields costs to the U.S. Healthcare System in billions of dollars per year. Chronic insomnia has been linked to numerous physical and psychological health outcomes as well as increased mortality.

There is also evidence that insomnia is a risk factor for worse inflammation, worse neurological functioning, cognitive performance, and mild cognitive impairment, including cognitive decline, Alzheimer's disease, and faster genetic and brain aging. Moreover, in patients with Alzheimer's disease those with insomnia showed a faster progression to dementia. Better sleep health provides neuroprotection against this decline. Impairment in objective and subjective cognitive performance, highlights the utility of treating insomnia to potentially improve cognitive outcomes during midlife and insomnia symptoms are a modifiable risk factor for cognitive decline, mild cognitive impairment, and Alzheimer's disease and related dementia.

Cognitive Behavioral Therapy for Insomnia (CBTi) is the gold-standard, first line recommended treatment for insomnia, and has considerably better long-term outcomes than medications. CBTi decreases insomnia symptom severity by 50%. CBTi also appears to improve cognitive functioning. However, CBTi is underutilized, training is limited, and medical professionals are implementing treatment approaches inconsistent with empirically supported guidelines. Insomnia symptoms are being inadequately treated while misinformation and misconceptions about insomnia disorder, CBTi, and actual therapeutic effects are being propagated. Moreover, sedating medications are currently the most commonly used treatment for insomnia, which is problematic because the potential side effects can have major implications for the aging population. Additionally, some patients continue to experience insomnia symptoms even when taking sleep medication, which can lead to increase dosages, dependence on, and tolerance to these medications, further emphasizing the importance of CBTi. There is also a need for more readily accessible, short-term, modified treatments for insomnia disorder. A modified format of CBTi may assist in dissemination of effective treatments while also providing the potential for adapting this treatment to specific client characteristics. To address this need, we will modify CBTi and conduct a pilot randomized clinical trial to test these modifications.

The proposed project will include two primary aims in establishing a foundation needed to examine individual benefits of the components of CBTi. These aims will aid in the continuation of investigation to better assess treatment outcomes, create transdiagnostic treatment plans, and provide individualized health care through accessible psychotherapy. Obtaining a better understanding of the predictors of successful treatment may improve our understanding of the underlying mechanisms of successful treatment. Ultimately, this improved understanding may help to improve treatment for insomnia disorder, improve cognitive functioning, and potentially reduced risk for cognitive decline associated with mild cognitive impairment, Alzheimer's disease, and related dementias. Improved treatment outcomes utilizing specific core components of CBTi may result in improvements of insomnia disorder and cognitive functioning and would provide a major step forward in understanding the mechanisms underlying the etiology and maintenance of insomnia as well as how risks associated with mild cognitive impairment and cognitive decline might be mitigated. Lastly, this proposed project allows for proof of concept and for collaborations to be made within the medical and mental health communities in Pocatello, ID and surrounding areas, decreasing barriers to treatment and improving treatment dissemination.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Seeking treatment for an insomnia complaint, assessed by self-report;
* Stable on any prescribed, non-sedating medications (≥ 1 month), assessed by self-report and structured clinical interview

Exclusion Criteria:

* Inability to speak and read English;
* Moderate to severe brain damage, assessed by the MoCA;
* Inability to attend weekly therapy sessions either in-person or via telehealth;
* Pregnancy, assessed by self-report, because sleep disturbances due to pregnancy may be the result of different processes;
* Other untreated sleep disorders (e.g., sleep apnea, periodic limb movement disorder), assessed by clinical interview. Participants meeting criteria for a sleep disorder requiring intervention will be referred for care through the local Medical Centers or their preferred sleep disorders center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | Baseline, Week 8, 1 Month Follow Up
  Sleep efficiency represents a ratio of total sleep time and total time in bed. Measured 0-100% with higher percentages indicating better sleep efficiency.
Insomnia Severity | Baseline, Weeks 1-6 of treatment, Week 8, 1 Month Follow Up
  Insomnia severity measured by the Insomnia Severity Index. Measured 0-28 with higher scores indicating worse insomnia severity.
Multidimensional Sleep Health | Baseline, Weeks 1-6 of treatment, Week 8, 1 Month Follow Up
  RU-SATED will be used to assess sleep health among adults. Measured 0-12 with higher scores indicating better sleep health.

SECONDARY OUTCOMES:
Cognitive Functioning | Baseline, Week 8
  Cognitive functioning will be assess with Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (EXAMINER). Measured by domain via T-Score.

OTHER OUTCOMES:
Improvements in Subjective Sleep | Baseline, Weeks 1-6 of treatment, Week 8, 1 Month Follow Up
  Subjective sleep will be assessed using a daily sleep diary.
Improvements in Objective Sleep | Baseline, Week 8
  Objective sleep will be measured with EEG and/or actigraphy.
Treatment Adherence and Attendance | Weeks 1-6 of treatment
  Treatment adherence will be assess by the clinician based on how closely and consistently the participants complete aspects of therapy. Attendance will be calculated by number of sessions attended.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Emert, Principal Investigator — Idaho State University
Locations (1):
- Idaho State University Psychology Clinic, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study data will be used for additional grant proposals.